CLINICAL TRIAL: NCT05399394
Title: Induction FOLFIRINOX Followed by Chemoradiation in Locally Advanced Pancreatic Cancer
Acronym: FOLRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000696-25
Record Dates: First submitted 2022-04-06; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer
Keywords: chemoradiation; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Neoadjuvant Therapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LAPC patients (Experimental): Patients treated with induction FOLFIRINOX; for patients without disease progression as detected through restaging exams, chemotherapy was followed by chemoradiation which consisted of conformal radiation therapy and concurrent gemcitabine at the dose of 600 mg/mq weekly.
  Interventions: Drug: Chemotherapy; Radiation: Radiation

INTERVENTIONS:
Drug: Chemotherapy — The induction phase of the treatment plan was designed to administer FOLFIRINOX protocol (oxaliplatin 85 mg/mq and irinotecan 180 mg/mq plus leucovorin 400 mg/mq followed by bolus fluorouracil (FU) 400 mg/mq on day 1, then FU 2,400 mg/mq as a 46-hour continuous infusion) every 14 days for four cycles. In the combined phase, concurrent chemotherapy consisted of weekly gemcitabine at the dose of 600 mg/mq.
  Other Names: Induction therapy
Radiation: Radiation — Radiotherapy target volumes are established by CT scan and PET-CT scan. Radiotherapy is delivered with a total dose of 54-59 Gy with fractionation of 1.8 Gy daily for 5 days a week. The Planning Target Volume (PTV) is defined by the Clinical Target Volume (CTV) with a safety margin to include organ motion and set-up errors. Organs at risk for radiation-induced side effects are contoured on the dose planning CT and dose volume histograms (DVH) are calculated. All treatments are delivered with a multifield isocentric technique using a multileaf collimator. A quality-control protocol are applied through cone-beam computed tomography systems (CBCT) for all patients to evaluate the precision of the set-up.

SUMMARY:
There is no a clear consensus regarding the optimal treatment strategy of locally advanced pancreatic cancer. There is a potential role for neoadjuvant therapy to treat micrometastatic disease with chemotherapy, as well as for the treatment of local disease with radiotherapy. The investigators evaluated the safety and efficacy of induction FOLFIRINOX followed by a high weekly dose of gemcitabine concurrent to radiation therapy in patients with borderline resectable and unresectable locally advanced pancreatic cancer (LAPC).

DETAILED DESCRIPTION:
Continued optimization in multimodality therapy and an accurate patient selection remain crucial points for the appropriate treatment of patients with pancreatic cancer. In all patients an accurate pre-treatment staging was performed, including multilayer CT scan, positron emission computed tomography (PET-CT) with 18F-2-fluoro-2-deoxy-D-glucose (FDG) and laparoscopy with peritoneal washing. Patients with the evidence of metastatic disease were excluded, and thus only a small number of patients was consequently enrolled with this approach.The induction phase of the treatment plan was designed to administer FOLFIRINOX protocol (oxaliplatin 85 mg/mq and irinotecan 180 mg/mq plus leucovorin 400 mg/mq followed by bolus FU 400 mg/mq on day 1, then FU 2,400 mg/mq as a 46-hour continuous infusion) every 14 days for four cycles. In the combined phase of the treatment radiotherapy target volumes were established by CT scan and PET-CT scan. Concurrent chemotherapy consisted of gemcitabine at the dose of 600 mg/mq weekly. Four weeks after the completion of radiochemotherapy, restaging including CT scan and PET-CT scan was performed. Tumor response was defined in accordance with the World Health Organization (WHO) definition through CT scan and PET-CT scan. Surgery was considered in patients whose tumors were technically resectable. After resection, patients were evaluated every three months by means of a standard surveillance protocol that included history and physical examination, cross-sectional imaging and measurement of serum markers, and the intervals were extended to six months after two years

ELIGIBILITY:
Inclusion Criteria:

* proven cytological or histological diagnosis of pancreatic ductal adenocarcinoma;
* borderline resectable or unresectable pancreatic tumours;
* no previous radiochemotherapy to abdomen;
* 0-I Eastern Cooperative Oncology Group (ECOG) performance status;
* adequate cardiac, liver and kidney function and a good bone marrow reserve.

Exclusion Criteria:

* resectable and metastatic disease;
* previous or concomitant malignant disease;
* one or more of the following clinical conditions: infection, pregnancy or breast-feeding, liver failure, kidney failure, Pa O2 < 65 mmHg, Pa carbon dioxide (CO2) > 40 mmHg, mental disability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | four months
  During treatment, patients are evaluated through a directed history, weekly physical examination and blood exams. The occurrence and nature of any adverse events are recorded in accordance with the National Cancer Institute Common Toxicity Criteria (version 4.02) scale. When multiple treatment-related adverse events of the same type occurred in the same patient, only the most severe ones are reported. Subsequently, the dose of chemotherapy is adjusted according to the number of occurrences of grade 2 or greater events.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Overall Survival (OS) is determined from the day of the histological diagnosis. OS curves are calculated with the Kaplan-Meier method.
Progression-free survival | 3 years
  Progression-free survival (PFS) is obtained from the beginning of treatment to the observation of progression/recurrence, or to last follow-up if no event is observed. PFS curves are calculated with the Kaplan-Meier method.
Metastases-free survival | 3 years
  Metastases-free survival (MFS) is obtained from the beginning of treatment to the observation of distant progression, or to last follow-up if no event is observed. MFS curves are calculated with the Kaplan-Meier method.
Incidence of Local-regional Tumor Control | 3 years
  Patients are not considered to have local-regional control unless they achieve at least a partial response of their primary tumor or stable disease by imaging. Patients who do not achieve objective response are considered to have local-regional failure. Local-regional control rates are analyzed using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Fiore, MD, Principal Investigator — Campus Bio-Medico University

IPD SHARING:
Plan to Share IPD: No